CLINICAL TRIAL: NCT02088008
Title: A Randomized, Open-label, Single Dosing, Two-way Crossover Clinical Trial to Compare the Safety/Tolerability and Pharmacokinetics of the Combination of Cilnidipine 10mg and Valsartan 160mg in Comparison to Each Component Coadministered in Healthy Male Volunteers
Brief Title: A Bioequivalence Study Comparing Cilnidipine/Valsartan Combination Tablet With Coadministration of Cilnidipine and Valsartan
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ID_IDCV_1303
Record Dates: First submitted 2014-03-10; First posted 2014-03-14 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- cilnidipine/valsartan (Experimental): cilnidipine/valsartan tablet
  Interventions: Drug: cinidipine, valsartan
- cilnidipine+valsartan (Active Comparator): coadministration of cilnidipine and valsartan
  Interventions: Drug: cinidipine, valsartan

INTERVENTIONS:
Drug: cinidipine, valsartan

SUMMARY:
A randomized, open-label, single dosing, two-way crossover clinical trial to compare the safety/tolerability and pharmacokinetics of the combination of Cilnidipine 10mg and Valsartan 160mg in comparison to each component coadministered in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 40
* Signed informed consent

Exclusion Criteria:

* Has a history of hypersensitivity to IP ingredients
* Hypertension or hyportension

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2014-05; Primary Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
AUClast | 0~24hrs
Cmax | 0~24hrs

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea